CLINICAL TRIAL: NCT00633269
Title: Open, Non-Randomized, Single Centre Phase I Study to Assess the Metabolism, Excretion and Pharmacokinetics of a Single Oral 100 mg Dose of [14C]-AZD2281 (KU-0059436) in Patients With Advanced or Metastatic Solid Tumours Refractory to Standard Treatments
Brief Title: Study Assessing Metabolism, Excretion and Pharmacokinetics of a Poly (ADP-Ribose) Polymerase (PARP) Inhibitor in Patients With Solid Metastatic Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: KuDOS Pharmaceuticals Limited (Industry)
Responsible Party: Jim Carmichael - CMO, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0810C00010; KU36-37
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Neoplasm Metastasis
Keywords: Poly(ADP ribose) polymerases; Metastatic Solid Tumours
MeSH Terms: conditions — Neoplasm Metastasis | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD2281 — 100mg Oral Dose
  Other Names: Olaparib

SUMMARY:
Open, non-randomized, radiolabelled, single centre study designed to characterize the metabolism, excretion and pharmacokinetics of a single oral dose of 100 mg [14C]-radiolabelled AZD2281 (KU-0059436) in patients with advanced or metastatic solid tumours.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic tumour, refractory to standard therapies

Exclusion Criteria:

* Anti-cancer therapy including chemotherapy, radiotherapy (excluding palliative radiotherapy), endocrine therapy, immunotherapy or use of other investigational agents within 4 weeks prior to study entry.
* Patients may continue the use of LHRH agonists for cancer, bisphosphonates for bone disease and corticosteroids provided the dose is stable before and during the study.
* Females will be able to continue to take hormone replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To characterize the metabolism, excretion and pharmacokinetics of a single oral dose of 100 mg [14C]-radiolabelled AZD2281 (KU-0059436) in patients with advanced or metastatic solid tumours, assessed by blood, urine and faecal sampling | Various timepoints

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of AZD2281 (KU-0059436) by assessment of adverse events, laboratory findings and vital signs.
To provide plasma and excreta samples for future studies to investigate metabolite profiles and characterize human metabolites
To make a preliminary evaluation of clinical response as measured by objective tumour response rates at various timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: James Carmichael, BSc, MBChB, MD, FRCP, Study Director — KuDOS Pharmaceuticals, Ltd; Johann deBono, MD, FRCP, MSc PhD, Principal Investigator — Royal Marsden Hospital, Surrey, UK
Locations (1):
- Research Site, London, United Kingdom